CLINICAL TRIAL: NCT06795581
Title: PET Imaging of Phosphodiesterase-4B (PDE4B) in Alcohol Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10002210; 002210-M
Record Dates: First submitted 2025-01-25; First posted 2025-01-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11-19

CONDITIONS: Alcohol Use Disorder
Keywords: PET Imaging; Alcohol Use Disorder (AUD); Phosphodiesterase-4B (PDE4B)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- One-arm (Other): All subjects will receive the same tests.
  Interventions: Drug: 18F-PF-06445974

INTERVENTIONS:
Drug: 18F-PF-06445974 — Injected IV followed by PET scanning

SUMMARY:
Background:

People with alcohol use disorder (AUD) also often have bouts of depression called major depressive episodes (MDEs). People having MDEs have been found to have low levels of a protein called PDE4B in the brain. Researchers want to find out if people with AUD also have low levels of PDE4B. This research may help lead to better treatments for AUD.

Objective:

To find out (1) if PDE4B levels are lower in people who are withdrawing from AUD and (2) if their PDE4B levels go up after they abstain from alcohol for 3 to 4 weeks.

Eligibility:

Adults aged 18 to 70 years with AUD. They must be enrolled in protocol 14-AA-0181.

Design:

Participants enrolled in protocol 14-AA-0181 will stay in the clinic for 3 to 4 weeks for alcohol withdrawal. During this stay, they will have some added procedures for the current study.

Within the first week, participants will have a positron emission tomography (PET) scan of the brain. A needle will be used to guide a thin plastic tube (catheter) into a vein in one arm. An experimental substance called a radioactive tracer will be injected through the catheter. This tracer binds to PDE4B and makes it easier to see the protein in the brain. For the scan, participants will lie on a table that slides into a doughnut-shaped machine.

Participants will have a second PET scan toward the end of their stay in the clinic.

Participants may also have a magnetic resonance imaging (MRI) scan of the brain. They will lie on a bed that slides into a tube....

DETAILED DESCRIPTION:
Study Description:

AUD participants will be referred from protocol 14-AA-0181, which includes a four-week hospitalization at NIH for alcohol withdrawal. Using the PET radioligand [18F]PF974 to measure the density of PDE4B, AUD participants will be scanned twice: 1) within one week of admission, and 2) after 3-4 weeks of alcohol withdrawal.

Objectives:

Primary Objective #1: To determine whether PDE4B radioligand binding is decreased in AUD participants during acute withdrawal compared to healthy volunteers matched as a group for age and sex.

Primary Objective #2: To determine whether PDE4B radioligand binding increases in individuals on the second scan compared to the first.

Secondary Objective: No exploratory correlations are hypothesized for this novel imaging of PDE4B. However, we may later perform correlations with any of the clinical parameters or biological biomarkers obtained in the 14- AA-0181. Note that Dr. Diazgranados is an AI of this PET protocol, and Dr. Innis will become an AI of the parent protocol.

Endpoints:

Primary endpoint: For both objectives, the primary endpoint is PET measurement of PDE4B binding (VT) in all regions of the brain.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18-70 years
  2. Willingness to complete the study including MRI tests.
  3. Each participant must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
  4. Participants must have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
  5. Participants must agree to adhere to the lifestyle considerations.
  6. Enrolled in protocol 14-AA-0181

EXCLUSION CRITERIA:

Clinically significant abnormalities on laboratory testing beyond that expected in participants during alcohol withdrawal. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen).

1. Clinically significant abnormalities on EKG.
2. Participants who, in the investigator s judgment, pose a current serious suicidal or homicidal risk.
3. Participants with a breath alcohol level (BAL) past 0.08.
4. Participants who have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
5. Participants who have taken antidepressants or antipsychotic medications in the week prior or during their hospital admission.
6. HIV infection.
7. Pregnancy.
8. Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
9. Have an inability to lie flat and/or lie still on the camera bed for two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the participant during the screening visit.
10. Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.
11. Be NIMH staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2028-12-11 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
To measure distribution volume | 36 months
  Target quantification

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The results will be submitted to ClinicalTrials.gov@@@@@@
Supporting Information: Study Protocol
Time Frame: 18 months after closure of protocol@@@@@@
Access Criteria: BTRIS

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002210-M.html